CLINICAL TRIAL: NCT00936104
Title: Prognostic and Therapeutic Relevance of the 'Side Population' in Pancreatic Cancer
Brief Title: Side Population in Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Baki Topal, Professor of Surgery, University Hospital, Gasthuisberg
Other Study IDs: BT-PDAC-SP
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Neoplasm; Pancreas
Keywords: pancreas; cancer; stem cell
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pancreatic cancer tissue specimen

GROUPS / COHORTS (1):
- SP in PDAC: Side population cells isolated from resection specimens obtained from patients with pancreatic cancer

SUMMARY:
In the current project we aim to study the oncological process of pancreatic cancer, from a perspective of the CSC-theory and in particular through the 'side population' (SP)-approach. The SP seems to be enriched for CSC and doesn't a priori exclude any CSC-subpopulation. After isolation from pancreatic cancer resection specimens, SP cells will be characterized by gene-expression profiling based on microarray analysis. We'll identify markers and pathways (with emphasis for stem cell and cancer -related ones) that are differentially expressed in SP versus the rest of tumour cells (the 'main population' or MP). In order to assess the prognostic relevance of the SP, we'll study these genes using the high-throughput Nanostring technology in about 200 snap-frozen PDAC resection specimens of patients from our prospective database. Finally, two monoclonal antibodies (mAB) will be tested as novel therapeutic agents in vivo (mouse model), wherein the choice of mAB will be based on prognostically relevant molecular targets and pathways obtained from the Nanostring results.

ELIGIBILITY:
Inclusion Criteria:

* Resected pancreatic ductal adenocarcinoma (PDAC)
* Informed consent

Exclusion Criteria:

* Age < 18years
* Pregnancy
* Pre-operative radiotherapy
* Pre-operative chemotherapy
* IPMT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SP cells will be identified through incubation with vital dye Hoechst 33342 of cell suspensions that are obtained from fresh human pancreatic cancer resection specimens.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Characterization of side population (SP) cells in pancreatic ductal adenocarcinoma (PDAC)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Van den Broeck A, Gremeaux L, Topal B, Vankelecom H. Human pancreatic adenocarcinoma contains a side population resistant to gemcitabine. BMC Cancer. 2012 Aug 15;12:354. doi: 10.1186/1471-2407-12-354. PMID 22894607